CLINICAL TRIAL: NCT02885753
Title: Systemic Oxaliplatin or Intra-arterial Chemotherapy Combined With LV5FU2 +/- Irinotecan and an Target Therapy in First Line Treatment of Metastatic Colorectal Cancer Restricted to the Liver
Acronym: OSCAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 49
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal; cancer; metastasis; hepatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Leucovorin; Oxaliplatin; Panitumumab; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Experimental arm FOLFOX with oxaliplatin intraarterial + targeted therapy to RAS status (Experimental): Panitumumab (6 mg/kg if RAS wild) or Bevacizumab (5 mg/Kg if RAS mutated) Oxaliplatin (85 mg/m²) intraarterially Folinic Acid (400 mg/m²) intravenously 5Fu: 400 mg/m² in bolus of 10 minutes 5Fu: 2400 mg/m² intravenously over 46 hours
  Interventions: Drug: 5 FU bolus; Drug: Folinic acid; Drug: Oxaliplatin intra-arteriel; Drug: Panitumumab; Drug: Bevacizumab; Drug: 5 FU continuous
- Reference arm FOLFOX with oxaliplatin intravenous + targeted therapy to RAS status (Active Comparator): Panitumumab (6 mg/kg if RAS wild) or Bevacizumab (5 mg/Kg if RAS mutated) Oxaliplatin (85 mg/m²) intravenously Folinic Acid (400 mg/m²) intravenously 5Fu: 400 mg/m² in bolus of 10 minutes 5Fu: 2400 mg/m² intravenously over 46 hours
  Interventions: Drug: Oxaliplatin intravenous; Drug: 5 FU bolus; Drug: Folinic acid; Drug: Panitumumab; Drug: Bevacizumab; Drug: 5 FU continuous
- Experimental arm mFOLFIRINOX with oxaliplatin intraarterial + Bevacizumab (Experimental): Bevacizumab (5 mg/Kg) Oxaliplatin (85 mg/m²) intraarterially Irinotecan (150 mg/m²) intravenously Folinic Acid (400 mg/m²) intravenously 5Fu: 2400 mg/m² intravenously over 46 hours
  Interventions: Drug: Folinic acid; Drug: Oxaliplatin intra-arteriel; Drug: Bevacizumab; Drug: 5 FU continuous; Drug: Irinotecan
- Reference arm mFOLFIRINOX with oxaliplatin intravenous + Bevacizumab (Active Comparator): Bevacizumab (5 mg/Kg) Oxaliplatin (85 mg/m²) intravenously Irinotecan (150 mg/m²) intravenously Folinic Acid (400 mg/m²) intravenously 5Fu: 2400 mg/m² intravenously over 46 hours
  Interventions: Drug: Oxaliplatin intravenous; Drug: Folinic acid; Drug: Bevacizumab; Drug: 5 FU continuous; Drug: Irinotecan

INTERVENTIONS:
Drug: Oxaliplatin intravenous — 85 mg/m² in intravenous. 1 cycle each 15 days
  Other Names: Oxaliplatin IV
  Arms: Reference arm FOLFOX with oxaliplatin intravenous + targeted therapy to RAS status; Reference arm mFOLFIRINOX with oxaliplatin intravenous + Bevacizumab
Drug: 5 FU bolus — 5 fluorouracil : 400 mg/m² in bolus of 10 minutes (intravenous) following by 2400 mg/m² during 46 hours in intravenous
  Other Names: 5 FU
  Arms: Experimental arm FOLFOX with oxaliplatin intraarterial + targeted therapy to RAS status; Reference arm FOLFOX with oxaliplatin intravenous + targeted therapy to RAS status
Drug: Folinic acid — 400 mg/m² in intravenous
  Other Names: Folinic Acid IV
Drug: Oxaliplatin intra-arteriel — 85 mg/m² in intra-arterial. 1 cycle each 15 days
  Other Names: Oxaliplatin IA
  Arms: Experimental arm FOLFOX with oxaliplatin intraarterial + targeted therapy to RAS status; Experimental arm mFOLFIRINOX with oxaliplatin intraarterial + Bevacizumab
Drug: Panitumumab — Only for patient RAS wild: 6 mg/Kg at each cycle in intravenous
  Other Names: Pani
  Arms: Experimental arm FOLFOX with oxaliplatin intraarterial + targeted therapy to RAS status; Reference arm FOLFOX with oxaliplatin intravenous + targeted therapy to RAS status
Drug: Bevacizumab — 5 mg/kg at each cycle in intravenous
  Other Names: Beva
Drug: 5 FU continuous — 2400 mg/m² intravenously over 46 hours
  Other Names: 5 FU
Drug: Irinotecan — 150 mg/m² intravenous
  Other Names: IRI
  Arms: Experimental arm mFOLFIRINOX with oxaliplatin intraarterial + Bevacizumab; Reference arm mFOLFIRINOX with oxaliplatin intravenous + Bevacizumab

SUMMARY:
Colorectal cancer is the 3rd most common cancer in France and the 2nd cause of death from cancer. Between 30 to 60% of patients develop limited or predominant liver metastases. Surgical resection of these metastases, only curative treatment is not immediately possible in 10-15% of cases. In unresectable patients, current palliative treatments are based on systemic chemotherapy associated or not with the targeted therapies (anti-EGFR (panitumumab), anti-VEGF (bevacizumab)). In this patient population, special attention was paid to intensified treatment regimens in order to improve their efficiency and improving the tumoral response rate, the intensity of the response and its earliness correlate with improved overall and progression-free survival.

The intra-arterial use of oxaliplatin coupled with IV chemotherapy has yielded OR levels of 64% in patients having survived one or more lines of chemotherapy IV and 62% in patients who have progressed on oxaliplatin IV. In addition, the HIA administration of oxaliplatin limits systemic and especially neurological toxicities, thanks to a greater hepatic clearance.

In conclusion, the combination of systemic chemotherapy, targeted therapy and HIAC with oxaliplatin has showed promising efficacy results associated with good tolerance from the first line onwards. Indeed, we can expect from the Phase II recent data, a control rate close to 100%, with high response rates associated with early maturity and depth responses as well as prolonged survival. However, to date, in the absence of randomized trial testing this combination, this strategy does not have sufficient evidence to be integrated in our routine practices, and HIAC remains limited to a few expert centers in treatment catch-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma with hepatic metastasis(es)
* At least one measurable hepatic metastasis according to the criteria RECIST v1.1
* No other metastatic sites except lung nodules if number ≤ 3 and < 10 mm
* RAS mutation status known (determination of KRAS mutation (exons 2,3 and 4) and determination of the NRAS mutation (exons 2,3 and 4))
* Age ≥ 18
* WHO ≤ 2 (Appendix 4)
* No prior treatment by chemotherapy except perioperative or adjuvant chemotherapy discontinued for more than 12 months
* Life expectancy > 3 months
* PNN > 1500/mm3, platelets > 100 000/mm3, Hb > 9 g/dLq
* Bilirubin < 25 mmol/L, AST < 5x ULN, ALT < 5 x ULN, ALP < 5 x ULN, TP > 60%, proteinuria from 24H < 1 g
* Creatinine clearance > 50 mL/min according to MDRD formula (Appendix 4)
* Patient affiliated to a social security scheme
* Patient information and signature of the informed consent

Exclusion Criteria:

* Contraindications specific to the installation of a KTHIA: thrombosis of the hepatic artery, arterial vascular anatomy may compromise a secondary hepatic resection.
* Patient immediately eligible for a curative therapy (surgical and/or percutaneous) after discussion in CPR
* Following alterations in the 6 months prior to inclusion: myocardial infarction, angina, severe/unstable angina, coronary artery bypass surgery, congestive heart failure NYHA class II, III or IV, stroke or transient ischemic attack
* Hypertension not controlled by medical treatment (SBP > 140 mmHg and/or DBP> 90 mmHg with blood pressure taken according to the diagram of the HAS)
* A history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active gastrointestinal bleeding in the 6 months preceding the start of treatment
* Progressive gastroduodenal ulcer, wound or fractured bone
* Abdominal or major extra-abdominal surgery (except diagnostic biopsy) or irradiation in the 4 weeks before starting the treatment
* Transplant patients, HIV positive or other immune deficiency syndromes
* Any progressive pathology not balanced over the past 6 months: hepatic failure, renal failure, respiratory failure
* Peripheral neuropathy > 1
* Patient with interstitial pneumonitis or pulmonary fibrosis
* History of chronic diarrhea or inflammatory disease of the colon or rectum, or unresolved occlusion or sub-occlusion in symptomatic treatment
* History of malignant pathologies during the past 5 years except basocellular skin carcinoma considered in complete remission or in situ cervical carcinoma, properly treated
* Patient already included in another clinical trial with an experimental molecule
* Any known specific contraindication or allergy or hypersensitivity to the drugs used in the study (cf RCP Appendix 7)
* Known deficit in DPD
* QT/QTc range > 450 msec for men and > 470 msec for women
* K+ < LNL, Mg2+ < LNL, Ca2+ < LNL
* Lack of effective contraception in patients (men and/or women) of childbearing age, pregnant or breastfeeding women, women of childbearing age not having had a pregnancy test
* Persons deprived of liberty or under supervision
* Impossibility of undergoing medical monitoring during the trial for geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 24 months after randomization
  comparison of radiological/clinical progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Julien TAIEB, MD-PhD, Principal Investigator — HEGP, Paris
Locations (49):
- Hôpital Erasme, Brussels, Belgium
- France (48):
  - Chu Hotel Dieu, Angers
  - Institut de Cancérologie de l'Ouest, Angers
  - Hôpital Privé d'Antony, Antony
  - CH Henri Duffaut, Avignon
  - Institut du cancer Avignon Provence, Avignon
  - Ch Cote Basque, Bayonne
  - Clinique Belharra, Bayonne
  - Centre Hospitalier, Beauvais
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - CH Loire Vendée Océan, Challans
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Chu Le Bocage, Dijon
  - Chd Vendee, La Roche-sur-Yon
  - Groupe Hospitalier de la Rochelle Re-Aunis, La Rochelle
  - Ch de Bicetre, Le Kremlin-Bicêtre
  - GH Nord Essone, Longjumeau
  - Hôpital du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Européen, Marseille
  - Hôpital Saint-Joseph, Marseille
  - Institut Paoli Calmettes, Marseille
  - Chu Hotel Dieu, Nantes
  - CHR La Source, Orléans
  - Hôpital Cochin, Paris
  - Hôpital Saint Joseph, Paris
  - Hôpital Saint Louis, Paris
  - Paris Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier, Pau
  - Centre Hospitalier Saint Jean, Perpignan
  - CHU Haut Lévêque, Pessac
  - CHU La Milétrie, Poitiers
  - Centre Eugène Marquis, Rennes
  - Clinique Pasteur, Ris-Orangis
  - CROME, Ris-Orangis
  - CHU Charles Nicolle, Rouen
  - CHP, Saint-Grégoire
  - Institut de cancérologie de l'Ouest, Saint-Herblain
  - CHU Saint-Etienne, Saint-Priest-en-Jarez
  - Hôpital FOCH, Suresnes
  - Maison de Santé Protestante de Bordeaux Bagatelle, Talence
  - Hia Sainte Anne, Toulon
  - Chu Toulouse Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
  - Hôpital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pernot S, Pellerin O, Mineur L, Monterymard C, Smith D, Lapuyade B, Gallois C, Khemissa Akouz F, De Baere T, Tougeron D, Thirot-Bidault A, Audemar F, Simon M, Lecaille C, Louafi S, Lepage C, Ducreux M, Taieb J. Phase III randomized trial comparing systemic versus intra-arterial oxaliplatin, combined with LV5FU2 +/- irinotecan and a targeted therapy, in the first-line treatment of metastatic colorectal cancer restricted to the liver (OSCAR): PRODIGE 49. Dig Liver Dis. 2022 Mar;54(3):324-330. doi: 10.1016/j.dld.2021.12.012. Epub 2022 Jan 11. PMID 35027324